CLINICAL TRIAL: NCT02511405
Title: A Phase 3, Randomized, Controlled, Double-Arm, Open-Label, Multi-center Study of VB-111 Combined With Bevacizumab vs. Bevacizumab Monotherapy in Patients With Recurrent Glioblastoma
Brief Title: A Phase 3, Pivotal Trial of VB-111 Plus Bevacizumab vs. Bevacizumab in Patients With Recurrent Glioblastoma (GLOBE)
Acronym: GLOBE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VB-111-215
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2017-01

CONDITIONS: Glioblastoma
Keywords: rGBM; Recurrent Glioblastoma; Recurrent GBM
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): VB-111 + Bevacizumab
  Interventions: Drug: VB-111 + bevacizumab
- Arm 2 (Active Comparator): Bevacizumab
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: VB-111 + bevacizumab — VB-111 will be administered intravenously at a dose of 1x10e13 VPs every 2 months
  Bevacizumab will be administered intravenously at a dose of 10mg/kg every 2 weeks
  Arms: Arm 1
Drug: Bevacizumab — Bevacizumab will be administered intravenously at a dose of 10mg/kg every 2 weeks
  Arms: Arm 2

SUMMARY:
The purpose of this pivotal, phase 3, randomized, multicenter study is to compare VB-111 plus bevacizumab to bevacizumab in adult patients with recurrent Glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. First or second progression of Glioblastoma;
2. Measurable disease by RANO criteria at progression;
3. Patients ≥18 years of age;
4. Patient may have been operated for recurrence. If operated: residual and measurable disease after surgery is required;
5. Surgery completed at least 28 days before randomization;
6. An interval of at least 12 weeks between prior radiotherapy or at least 23 days from prior chemotherapy, 42 days from nitrosoureas and enrollment in this study;
7. Adequate performance, i.e."Karnofsky Performance Score" of at least 70%;
8. Adequate renal, liver, and bone marrow function according to the following criteria:

   * Absolute neutrophil count ≥1500 cells/ml,
   * Platelets ≥ 100,000 cells/ml,
   * Total bilirubin within upper limit of normal (ULN),
   * Aspartate aminotransferase (AST) ≤ 2.0 X ULN,
   * Serum creatinine level ≤ ULN or creatinine clearance ≥ 50 ml/min for patients with creatinine levels above normal limits (creatinine clearance calculated by the Cockcroft-Gault formula, see Appendix II),
   * PT, PTT (in seconds) not to be prolonged beyond >20% of the upper limits of normal.

Exclusion Criteria:

1. Prior anti-angiogenic therapy including VEGF sequestering agents (i.e. bevacizumab, aflibercept, etc.) or VEGFR inhibitors (cedirinib, pazopanib, sunitinib, sorafenib, etc.);
2. Prior stereotactic radiotherapy;
3. Pregnant or breastfeeding patients;
4. Concomitant medication that may interfere with study results; e.g. immunosuppressive agents other than corticosteroids;
5. Active infection;
6. Evidence of significant CNS haemorrhage i.e. CTCAE grade 2 or above;
7. Expected to have surgery during study period;
8. Patients with active vascular disease, either myocardial or peripheral (i.e. acute coronary syndrome, cerebral stroke, transient ischemic attack or arterial thrombosis or symptomatic peripheral vascular disease within the past 3 months);
9. Patients with known proliferative and/or vascular retinopathy;
10. Patients with known liver disease (alcoholic, drug/toxin induced, genetic, or autoimmune);
11. Patients with known active second malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, and ductal or lobular carcinoma in situ of the breast. Patients are not considered to have a currently active malignancy if they have completed anticancer therapy and have been disease free for greater than 2 years prior to screening;
12. Patients testing positive to one of the following viruses: HIV, HBV and HCV within the last 6 months;
13. Patients that have undergone major surgery within the last 4 weeks before enrollment;
14. Patients who have received treatment with any other investigational agent within 4 weeks before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-11-03 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of study entry until the date of death from any cause (up to 10 years)

SECONDARY OUTCOMES:
Progression Free Survival | To be assessed from date of randomization until the date of disease progression, assessed up to 10 years.
Tumor response as measured by RANO Criteria | To be assessed from date of randomization until the date of disease progression, assessed up to 10 years.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (48):
  - University of Alabama, Birmingham, Alabama
  - Highlands Oncology Group, Rogers, Arizona
  - University of California Irvine Medical Center, Irvine, California
  - University of California Los Angeles, Los Angeles, California
  - The Center for Cancer Prevention and Treatment, Orangevale, California
  - Kaiser Permanente - Redwood City Medical Center, Redwood City, California
  - University of California, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Colorado Neurological Institute, Denver, Colorado
  - The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida Preston A. Wells, Jr. Center for Brain Tumor Therapy, Gainesville, Florida
  - Orlando Health, Orlando, Florida
  - Piedmont Physicians Neuro-Oncology, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Louisiana State University Health Science Center, Shreveport, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Metro-MN Community Oncology Research Consortium, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dent Neurosciences Research Center, Amherst, New York
  - North Shore University Hospital, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Derald H. Ruttenberg Treatment Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University, Neurology Associates of Stony Brook, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Baylor Health Neuro-Oncology Associates, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - : University of Texas, HSC, Houston, Texas
  - MD Anderson, Houston, Texas
  - UTHSCSA, San Antonio, Texas
  - Huntsman Cancer Institute at The University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petach Tikvah
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Ellingson BM, Hagiwara A, Morris CJ, Cho NS, Oshima S, Sanvito F, Oughourlian TC, Telesca D, Raymond C, Abrey LE, Garcia J, Aftab DT, Hessel C, Rachmilewitz Minei T, Harats D, Nathanson DA, Wen PY, Cloughesy TF. Depth of Radiographic Response and Time to Tumor Regrowth Predicts Overall Survival Following Anti-VEGF Therapy in Recurrent Glioblastoma. Clin Cancer Res. 2023 Oct 13;29(20):4186-4195. doi: 10.1158/1078-0432.CCR-23-1235. PMID 37540556
- [Derived] Cloughesy TF, Brenner A, de Groot JF, Butowski NA, Zach L, Campian JL, Ellingson BM, Freedman LS, Cohen YC, Lowenton-Spier N, Rachmilewitz Minei T, Fain Shmueli S; GLOBE Study Investigators; Wen PY. A randomized controlled phase III study of VB-111 combined with bevacizumab vs bevacizumab monotherapy in patients with recurrent glioblastoma (GLOBE). Neuro Oncol. 2020 May 15;22(5):705-717. doi: 10.1093/neuonc/noz232. PMID 31844890
- See also: VBL Therapeutics Company Website — http://www.vblrx.com